CLINICAL TRIAL: NCT03947996
Title: Comparison of Stretching and Walking as Exercise Modalities for Reducing Blood Pressure
Brief Title: Stretching Versus Walking From Reducing Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1133
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Parallel groups: Two groups: Walking exercise and stretching exercise
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching (Experimental): Stretching
  Interventions: Other: Stretching exercise
- Walking (Experimental): Walking
  Interventions: Other: Walking exercise

INTERVENTIONS:
Other: Stretching exercise — Stretching (30 minutes, 5 days per week, 8 weeks)
  Arms: Stretching
Other: Walking exercise — Walking (30 minutes, 5 days per week, 8 weeks)
  Arms: Walking

SUMMARY:
High blood pressure is a leading risk factor for cardiovascular disease. Traditionally, one of the ways to treat or prevent high blood pressure is to prescribe aerobic exercise training (i.e.brisk walking). Previous studies have shown that stretching is also very effective for reducing blood pressure. This is an exciting possibility because if stretching is more effective, it would change the way exercise is prescribed to people with elevated blood pressure. This study will now assess 20 individuals in a supervised stretching or walking program five days per week for 8 weeks to determine for certain whether stretching is superior for reducing blood pressure. This research will contribute to recommendations about the most effective exercise programs for reducing blood pressure and risk of cardiovascular disease.

DETAILED DESCRIPTION:
The study hypothesis is that stretching (flexibility training) will be superior to brisk walking for reducing blood pressure.

This is a parallel-group randomised trial. Twenty participants (aged 18 and older) with borderline or stage-1 hypertension (systolic blood pressure between 130 and 159 mmHg OR diastolic blood pressure between 85 and 99 mmHg) will be randomised to walking or stretching groups. Each group will do 30 minutes of exercise, five days per week. Exercise sessions will be supervised three days per week with participants doing exercise sessions on their own two days per week. Exercise sessions involve either brisk walking or stretching. The stretching exercises will involve stretching all major muscle groups. The main outcome is 24-hour blood pressure which will be assessed at baseline, after four weeks, and after eight weeks. Other outcomes will be assessed at baseline and eight weeks and include: Body weight, height, waist circumference, resting heart rate, physical activity levels (questionnaire), diet (questionnaire), maximal distance walked in six minutes. All participants will be counselled on how to follow the DASH eating plan, which involves reducing dietary salt intake.

Statistical analyses: All outcomes will be assessed with a group x time ANOVA with alpha level of 0.05. LSD post-hoc tests will be done when necessary to identify differences between pairs of means.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure between 130 and 159 mmHg OR diastolic blood pressure between 85 and 99 mmHg

Exclusion Criteria:

* Individuals will be excluded if they have taken blood pressure medications within the past six months unless they are on a stable dose of medication and have not reach target blood pressure levels (i.e. systolic blood pressure below 130 mmHg and diastolic blood pressure below 85 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Night time blood pressure | Change from Baseline Night Time Blood Pressure at 8 weeks
  Blood pressure assessed during the night with an automated device

SECONDARY OUTCOMES:
Day time blood pressure | Change from Baseline Day Time Blood Pressure at 8 weeks
  Blood pressure assessed during the day with an automated device
Sitting blood pressure | Change from Baseline Sitting Blood Pressure at 8 weeks
  Blood pressure assessed while sitting
Lying blood pressure | Change from Baseline Lying Blood Pressure at 8 weeks
  Blood pressure assessed while lying down
Walking test | Change from Baseline Walking Distance at 8 weeks
  Maximal distance walked in six minutes
Waist circumference | Change from Baseline Waist Circumference at 8 weeks
  Waist circumference measured with a measuring tape
Body mass | Change from Baseline Body Mass at 8 weeks
  Body mass measured with a scale
Resting heart rate | Change from Baseline Resting Heart Rate at 8 weeks
  Heart rate at rest measured with a heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ko J, Deprez D, Shaw K, Alcorn J, Hadjistavropoulos T, Tomczak C, Foulds H, Chilibeck PD. Stretching is Superior to Brisk Walking for Reducing Blood Pressure in People With High-Normal Blood Pressure or Stage I Hypertension. J Phys Act Health. 2021 Jan 1;18(1):21-28. doi: 10.1123/jpah.2020-0365. Epub 2020 Dec 18. PMID 33338988